CLINICAL TRIAL: NCT07042503
Title: Effects of Different Preoperative Oral Rehydration Protocols on Safety, Comfort, and Postoperative Outcomes in Elderly Patients Undergoing Thoracoscopic Radical Lung Cancer Surgery: A Randomized Controlled Trial
Brief Title: Effects of Different Preoperative Oral Rehydration Protocols in Undergoing Thoracoscopic Radical Lung Cancer Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: fish77033
Record Dates: First submitted 2025-06-16; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Delirium
Keywords: preoperative oral rehydration protocol; Postoperative delirium; insulin resistance; gastric emptying status; preoperative anxiety
MeSH Terms: conditions — Emergence Delirium; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control Arm: 2-hour Preoperative Ingestion of 200-300 mL clear water
- Intervention Arm 1: Hourly Preoperative Ingestion of 50-100 mL clear water
- Intervention Arm 2: Hourly Preoperative Ingestion of 50-100 mL 12.5% carbohydrate-containing beverages

SUMMARY:
This study aims to compare the new preoperative oral rehydration protocol (administering 50-100 mL of clear fluids or carbohydrate-rich beverages orally every hour until the patient arrives at the operating room) with the traditional preoperative protocol (consuming 200-300 mL of water orally two hours prior to surgery). The objective is to investigate the effects of these two protocols on the safety (e.g., risk of reflux and aspiration), comfort (e.g., levels of hunger, thirst, and anxiety), gastric emptying status (as assessed by gastric ultrasound indicators), and postoperative outcomes (e.g., incidence of postoperative delirium, insulin resistance, and inflammatory factor levels) in elderly patients undergoing thoracoscopic lung cancer radical surgery. This research seeks to identify a more appropriate preoperative rehydration protocol for elderly lung cancer patients.

DETAILED DESCRIPTION:
This study employed a randomized controlled double-blind trial, including 420 elderly patients (aged 65 and above) who were scheduled to undergo thoracoscopic lung cancer radical surgery. The efficacy of three preoperative oral rehydration regimens was compared. The control group orally consumed 200-300ml of clear water 2 hours before the operation; the intervention group 1 orally consumed 50-100ml of clear water every hour before the operation; the intervention group 2 orally consumed 50-100ml of 12.5% carbohydrate beverages every hour before the operation, all requiring to be consumed slowly within 10-15 minutes. The evaluation indicators included: safety (intraoperative reflux aspiration, postoperative nausea and vomiting, incision and pulmonary infection rates), gastric ultrasound (amount of fluid in the stomach and emptying time), comfort (VAS for assessing hunger and thirst, SAS for assessing anxiety), postoperative delirium (CAM scale combined with electroencephalogram), insulin resistance (FPG, FINS, and HOMA-IR), and inflammatory factors (Interleukin-6, Tumor necrosis factor -α, C-reactive protein). The research data were analyzed using SPSS software to clarify the impact of different rehydration regimens on elderly patients.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly patients aged 65 or above who are scheduled to undergo thoracoscopic radical lung cancer surgery.
2. American Society of Anesthesiologists (ASA) classification levels II-III.
3. No severe cognitive impairment (Mini-Mental State Examination (MMSE) score ≥ 24).
4. Able to cooperate with the study and sign the informed consent form.

Exclusion Criteria:

1. Combined with severe functional impairments of important organs such as the heart, liver, and kidneys.
2. Suffering from metabolic diseases such as diabetes and hyperthyroidism.
3. Having digestive system diseases such as gastric emptying disorders, dysphagia, and intestinal obstruction.
4. Allergic or intolerant to carbohydrates.
5. Had received treatments such as radiotherapy and chemotherapy before the surgery that might affect the research indicators.
6. Patients with mental disorders or cognitive dysfunction.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: elderly patients undergoing thoracoscopic lung cancer radical surgery
Sampling Method: Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
postoperative delirium | One to three days after the operation
  The Confusion Assessment Method - Short Form(CAM-S) scoring for postoperative delirium is as follows:
  Total score 20 points, 0-6 points :Mild delirium; 7-12 points:Moderate delirium;
  ≥13 points: Severe delirium.
preoperative anxiety | One day before the operation and in the morning of the operation
  The Generalized Anxiety Disorder-7 (GAD-7) scale for preoperative anxiety assessment is as follows:Total score: 21 points，0-4 points: Normal，5-9 points: Mild anxiety，10-14 points: Moderate anxiety，≥15 points: Severe anxiety.
The amount of fluid in the stomach | 2 hours before the operation, 1 hour before the operation, and before anesthesia induction
  Ultrasound examination of the cross-sectional area of the antrum of the stomach
insulin resistance | on the early morning of the day before the operation,the first day and the third day after operation
  venous blood was collected from the patients to detect fasting plasma glucose (FPG), insulin (FINS), and homeostasis model assessment of insulin resistance index (HOMA-IR).

SECONDARY OUTCOMES:
Perioperative hunger | 2 hours and 1 hour before the operation, before anesthesia induction and 6 hours after the operation
  The Visual Analogue Scale (VAS) allowed patients to rate their feelings of hunger (0-10 points, 0 for no hunger and 10 for extreme hunger) and thirst (0-10 points, 0 for no thirst and 10 for extreme thirst)
Perioperative thirst | 2 hours and 1 hour before the operation, before anesthesia induction and 6 hours after the operation
  The Visual Analogue Scale (VAS) was used to score the sensation of thirst (on a scale of 0 to 10, where 0 indicates no sensation of thirst and 10 indicates extreme thirst)
The incidence of reflux aspiration during the perioperative period | During the operation and 3 days after the operation
  Closely observe whether the patient has reflux or aspiration
The incidence of perioperative nausea and vomiting | During the operation and 3 days after the operation
  Record the frequency and severity of nausea and vomiting
C-reactive protein | on the early morning of the day before the operation,the first day and the third day after operation
  The fasting venous blood of the patients was collected and detected by immunoturbidimetry.
Tumor necrosis factor -α | on the early morning of the day before the operation,the first day and the third day after operation
  The fasting venous blood of the patients was collected and detected by enzyme-linked immunosorbent assay (ELISA).
Interleukin-6 | on the early morning of the day before the operation,the first day and the third day after operation
  The fasting venous blood of the patients was collected and detected by enzyme-linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Nan Lin, Principal Investigator — Fujian Medical University Union Hospital

IPD SHARING:
Plan to Share IPD: Undecided
The way of sharing IPD：ResMan, http://www.medresman.org.cn/login.aspx